CLINICAL TRIAL: NCT03150407
Title: A Pivotal Clinical Investigation to Evaluate the Safety and Efficacy of J3 Bioscience Lubricating Intravaginal Ring VR101 in Relieving Symptoms of Vaginal Dryness
Brief Title: Use of J3 Bioscience Lubricating Intravaginal Ring VR101 to Relieve the Symptoms of Vaginal Dryness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J3 Bioscience, Inc. (Industry)
Collaborators: Advanced Clinical Research Services, LLC (Other); Phil Triolo and Associates LC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CI02
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Results first posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Menopause Related Conditions; Postmenopausal Symptoms
Keywords: vaginal dryness; lubricant; lubrication; intravaginal ring; IVR; vaginal; extended release
MeSH Terms: interventions — Equipment and Supplies; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to GROUP V1S2 will insert a VR101 device and leave it in place for 7 days, then remove the first device and replace it with a fresh device on day 7. Subsequently, 2 additional devices will be inserted and removed serially on a 7-day schedule until a total of 4 devices are used by each study participant, with the last device removed at day 28.
  Participants assigned to S1V2 will insert a sham control ring and leave it in place for 7 days, then remove the first ring and replace it with a new ring on day 7. Subsequently, 2 additional sham rings will be inserted and removed serially on a 7-day schedule until a total of 4 sham rings are used by each study participant, with the last sham ring removed at day 28.
  Following completion of the first 28-day treatment course with either VR101 or sham control, participants will undergo a 21-day "washout" period during which no devices will be used, before "crossing over" to treatment with the other device.
Who Masked: Participant, Care Provider, Investigator
Masking Description: VR101 devices and Sham control rings differ only in that VR101 device rings contain glycerol-based lubricant, whereas the Sham controls do not. The product, either VR101 device or Sham ring, is randomly assigned to participants when they are enrolled in the study. Once inserted in the vagina, the devices are indistinguishable. Thus, Investigators cannot tell whether a VR101 device or Sham is in place while performing any vaginal examination. All products (VR101 devices or Sham rings) are intravaginally placed by participants in a room that is not occupied by Care Providers or Investigators, so it is impossible for them to know which product has been assigned. The packaging of all products is identical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- VR101 Device (Active Comparator): Subjects assigned to use randomly-assigned VR101 devices. Each device is to be used for 7 consecutive days, then replaced with a fresh device. Four each VR101 devices will be used. These will be investigated in a cross-over design that will also include consecutive use of 4 Shams, each for 7 days.
  Interventions: Device: VR101 Device (Efficacy)
- Sham Control Ring (Sham Comparator): Subjects assigned to use randomly-assigned Sham rings. Each Sham is to be used for 7 consecutive days, then replaced with a fresh sham. Four each Shams will be used. These will be investigated in a cross-over design that will also include consecutive use of 4 VR101 Devices, each for 7 days.
  Interventions: Other: Sham Control Ring
- Long-term Safety Evaluation (Other): 13-week investigation of the safety of the use of VR101 Devices
  Interventions: Device: VR101 Device (Safety)

INTERVENTIONS:
Device: VR101 Device (Efficacy) — Self-insertion of VR101 Device for 7 days, followed by replacement with a fresh VR101Device, until 4 each Devices have been used for 7 days each, with total consecutive device use equal to 28 days
  Other Names: VR 101; Device
  Arms: VR101 Device
Other: Sham Control Ring — Self-insertion of Sham Ring for 7 days, followed by replacement with a fresh Sham Ring, until 4 each Sham Rings have been used for 7 days each, with total consecutive Sham use equal to 28 days
  Other Names: Sham; Sham Ring; Control
  Arms: Sham Control Ring
Device: VR101 Device (Safety) — Following the 4-week use of shams and a 3-week washout period participants randomized to the Safety Study will use a new VR101 device every 7 days for 13 consecutive weeks.
  Other Names: VR 101; Device
  Arms: Long-term Safety Evaluation

SUMMARY:
This investigation is designed to demonstrate the safety and efficacy of the VR101 lubricating intravaginal ring (IVR) in treating the symptoms of vaginal dryness. In the proposed investigation, participants will use VR101 devices and sham control rings in a crossover study design. All participants who successfully complete the crossover study will be given the option to continue using VR101 for a total of 13 consecutive weeks to evaluate the long-term safety of the new device.

DETAILED DESCRIPTION:
CI02, A Pivotal Clinical Investigation to Evaluate the Safety and Efficacy of J3 Bioscience Lubricating Intravaginal Ring VR101 in Relieving Symptoms of Vaginal Dryness, is a multi-center, investigator- and participant-blind, randomized crossover study designed to evaluate the safety and efficacy of VR101 and establish its substantial equivalence to the predicate device, building on the results obtained in CI01, "VR101: A Pilot Study to Evaluate the Preliminary Feasibility and Safety of a Lubricating Intravaginal Ring to Relieve the Symptoms of Vaginal Dryness." The data from CI02 will be used to support a premarket 510(k) notification to the FDA to enable regulatory clearance of the device in the United States (US).

At least 60 participants (up to 69 may be enrolled to account for the anticipated drop-out rate) who consent to be enrolled and meet inclusion/exclusion criteria will be enrolled in the study. To qualify, women must be over the age of 35 who self-report having experienced vaginal dryness symptoms that interfere with daily activities, including but not limited to sexual activity, in the last 60 days; and their clinician-assigned baseline VHI score must be 22 or lower.

Enrolled participants will be randomly assigned to be treated initially by VR101 (GROUP V1S2) or a sham control (GROUP S1V2). Participants randomly assigned to GROUP V1S2 will insert a VR101 device and leave it in place for 7 days, then remove the first device and replace it with a fresh device on day 7. Subsequently, 2 additional devices will be inserted and removed serially on a 7-day schedule until a total of 4 devices are used by each study participant, with the last device removed at day 28.

Participants assigned to S1V2 will insert a sham control ring and leave it in place for 7 days, then remove the first ring and replace it with a new ring on day 7. Subsequently, 2 additional sham rings will be inserted and removed serially on a 7-day schedule until a total of 4 sham rings are used by each study participant, with the last sham ring removed at day 28.

Following completion of the first 28-day treatment course with either VR101 device or sham control, participants will undergo a 21-day "washout" period during which no products (devices or sham rings) will be used, before "crossing over" to treatment with the other product.

All participants who successfully complete the crossover study will be given the option to complete the long-term safety evaluation. V1S2 participants who elect to enter the safety study will switch back to VR101 following completion of the crossover study and use a new VR101 device every day for 13 consecutive weeks. S1V2 participants who elect to enter the safety study will continue using a new VR101 device every 7 days for 9 additional weeks, or a total of 13 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

Potential participants must:

* Completely understand and sign the informed consent form (ability to read and understand the consent form in the English language).
* Be female 35 years of age or older.
* Express willingness to comply with the study visit schedule (see Table 4 in study procedures section).
* Over the course of the study:

  * Express willingness to abstain from the use of any vaginal moisturizers or lubricants or any other topically applied vaginal products not provided by study staff during VR101 or sham use, or during the Washout Period
  * Express willingness to abstain from the use of any HRT (hormone replacement therapy) or hormone-containing birth control products
  * Express willingness to abstain from use of any vaginal ring, diaphragm, cervical cap, or pessary products
* In the previous 60 days, have self-reported vaginal dryness that interferes with daily activities, which may include sexual intercourse
* Present with a VHI score of 22 or less, as scored by a trained clinician during the initial visit

Exclusion Criteria:

Potential participants self-reporting any of the following will be ineligible for study entry:

* Current use of HRT (Hormone Replacement Therapy) or any hormone-containing birth control products.
* Vulvar or vaginal procedures (biopsies, radiation) in the last 3 months
* Active vulvar or vaginal infections/lesions or complaints, as well as undiagnosed abnormal genital bleeding
* History of chronic pelvic pain, interstitial cystitis, vulvar vestibulitis, pelvic inflammatory disease within the past 3 months
* Known current, clinically evident cervical or vaginal infection
* Participants who have given birth or terminated pregnancy in the past 6 weeks.
* Postpartum or post-abortion endometritis, unless symptoms resolved at least 3 months prior to study entry
* Current persistent, abnormal vaginal bleeding
* History of inability to place a vaginal ring
* History of any abnormality of the vagina resulting in distortion of the vaginal canal or incompatibility with intravaginal ring placement
* Body habitus or history of lower genital tract abnormalities or prior surgeries which may not allow the vagina to be appropriately accessed
* Known or suspected allergy or hypersensitivity to polyurethanes or glycerol
* Known current alcohol or illicit drug abuse
* Participants who have not recovered from adverse events due to chemotherapy or radiation treatment for cancer
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection of the urogenital tract, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any condition that in the opinion of the investigator or study staff that would constitute contraindications to participation in the study or would compromise ability to comply with the study protocol
* Current use of a vaginal ring, pessary, cervical cap or diaphragm unless willingness to discontinue for the study duration is expressed
* Pregnancy or plans to become pregnant in the next 6 months
* Current breastfeeding and inability or unwillingness to discontinue breastfeeding for the duration of the study

NOTE: IUD (Intrauterine Device, e.g., ParaGard®) users may be enrolled provided they commit to exercising caution when removing VR101 as IUD strings have been noted to interfere with VR101 removal.

NOTE: Participants who have previously undergone anterior and/or posterior vaginal repair and have received a vaginal mesh implant may have difficulty placing VR101, although no safety issues with VR101 use in CI01 participants who had vaginal mesh implants were noted.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must self-identify as female
Enrollment: 72 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Kirstein, MD, CPI, Principal Investigator — Advanced Clinical Research Services, LLC
Locations (2):
- United States (2):
  - Advanced Clinical Research, Inc. (ACR Idaho), Meridian, Idaho
  - Advanced Clinical Research, Inc. (ACR Utah), West Jordan, Utah

IPD SHARING:
Plan to Share IPD: No
There is no current plan to make individual patient data available to other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- V1S2: Participants randomly assigned to GROUP V1S2 were instructed to insert a VR101 device and leave it in place for 7 days, then remove the first device and replace it with a fresh device on day 7. Subsequently, participants were instructed to insert and remove 2 additional devices serially on a 7-day schedule until a total of 4 devices were used by each participant, with the last device removed at day 28.
  Following completion of the first 28-day treatment course with VR101, participants abstained from device use during a 21-day "washout" period before "crossing over" to use of the sham control for 4 weeks in an identical manner to that of VR101 use in the initial period. All participants who successfully completed both treatment periods were given the option to complete the long-term safety evaluation (13 additional weeks of VR101 use).
- S1V2: Participants assigned to S1V2 were instructed to insert a sham control ring and leave it in place for 7 days, then remove the first ring and replace it with a new ring on day 7. Subsequently, they were instructed to insert and remove 2 additional sham rings serially on a 7-day schedule until a total of 4 sham rings were used by each participant, with the last sham ring removed at day 28.
  Following completion of the first 28-day treatment course with the sham control, participants abstained from device use during a 21-day "washout" period before "crossing over" to use of VR101 for 4 weeks in an identical manner to that of sham control use in the initial period. All participants who successfully completed both treatment periods were given the option to complete the long-term safety evaluation (9 additional weeks of VR101 use, for a total of 13 consecutive weeks of VR101).
Period: Period 1
Arm/Group | V1S2 | S1V2
Started | 36 | 36
Completed | 32 | 34
Not Completed | 4 | 2
Period: Washout
Arm/Group | V1S2 | S1V2
Started | 32 | 34
Completed | 31 | 33
Not Completed | 1 | 1
Period: Period 2
Arm/Group | V1S2 | S1V2
Started | 31 | 33
Completed | 30 | 33
Not Completed | 1 | 0
Period: Long-Term Safety Extension
Arm/Group | V1S2 | S1V2
Started | 27 | 30
Completed | 26 | 27
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- V1S2: Participants randomly assigned to GROUP V1S2 were instructed to insert a VR101 device and leave it in place for 7 days, then remove the first device and replace it with a fresh device on day 7. Subsequently, participants were instructed to insert and remove 2 additional devices serially on a 7-day schedule until a total of 4 devices were used by each participant, with the last device removed at day 28.
- S1V2: Participants assigned to S1V2 were instructed to insert a sham control ring and leave it in place for 7 days, then remove the first ring and replace it with a new ring on day 7. Subsequently, they were instructed to insert and remove 2 additional sham rings serially on a 7-day schedule until a total of 4 sham rings were used by each participant, with the last sham ring removed at day 28.
- Total: Total of all reporting groups
Arm/Group | V1S2 | S1V2 | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (8.5) | 59.4 (8.5) | 59.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 31 | 34 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 35 | 35 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Menopausal Status [Count of Participants; unit: Participants] — During Visit 1, each participant was asked to report her menopausal status. Specifically, a participant was defined as menopausal if she had not experienced a menstrual period in the last 12 months.
  Participants
    Menopausal | 36 | 35 | 71
    Not Menopausal | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of VR101 Treatments at 28 Days Assessed by Change in VHI (Vaginal Health Index) Scores Assigned by Clinicians
Description: The Vaginal Health Index (VHI) ranges from 5 to 20 and is calculated via addition of clinician-determined ratings for Vaginal Elasticity, Fluid Volume, Epithelial Integrity, Moisture and pH (each ranges from 1 to 5, with 5 being the best).
Time Frame: Baseline, 28 Days
Population: "Completers Only": Participants that completed both study periods.
  "Worst-Case, Non-Statistical, Per-Protocol": Subjects who didn't complete a study period were assigned the last available score for Day 28. Subjects who missed an entire study period were assigned the worst-performing change score from the remaining population for Day 28.
  LOCF: Same as the per-protocol group, except participants missing an entire study period were assigned a change score of 0 (no efficacy) for that period.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- VR101: Combined 28-day composite VHI change scores during VR101 use across both groups / periods.
- Sham Control: Combined 28-day composite VHI change scores during sham control use across both groups / periods.
Arm/Group | VR101 | Sham Control
Number analyzed (Participants) | 72 | 72
Score on a Scale
  Completers Only: number analyzed (Participants) | 66 | 64
  Completers Only | 1.76 (3.32) | 0.55 (3.70)
  Worst-Case, Non-Statistical, Per-Protocol | 1.38 (3.55) | 0.97 (4.04)
  LOCF | 1.63 (3.21) | 0.49 (3.56)

2. Primary Outcome: Serious Adverse Device Effects
Description: Number of Participants with Serious Adverse Device Effects Over the VR101 Treatment Period
Time Frame: Up to 24 weeks total, comprising up to 17 weeks total VR101 use and up to 4 weeks total sham control use.
Measure: Count of Participants; unit: Participants
Groups:
- VR101: Participants with Serious Adverse Device Effects During VR101 Use
- Sham: Participants with Serious Adverse Device Effects During Sham Control Use
Arm/Group | VR101 | Sham
Number analyzed (Participants) | 72 | 72
Participants | 0 | 0

3. Other Pre Specified Outcome: Vaginal Dryness Severity Survey (Population Analysis)
Description: Claim 1: VR101 relieves the symptoms of vaginal dryness for up to 7 days.
  Participants were asked to rate the severity of their vaginal dryness on a four-point scale throughout the investigation. Responses were assigned numerical values as follows:
  * "I have not experienced vaginal dryness" (assigned a score of 0)
  * "Mild" (assigned a score of 1)
  * "Moderate" (assigned a score of 2)
  * "Severe" (assigned a score of 3)
  To assess the ability of VR101 to relieve the symptoms of dryness on the final day of ring use (nominally 7 days), participants were asked to report their dryness severity in the last 24 hours when removing their first VR101. This score was compared to the participant's assessment of their dryness severity in the week prior to VR101 use.
Time Frame: 7 Days
Population: Participants who completed their first week of VR101 use
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- VR101: Response measured after 1st week of VR101 use (across both groups)
- Baseline: Response measured before 1st week of VR101 use
Arm/Group | VR101 | Baseline
Number analyzed (Participants) | 66 | 66
Score on a Scale | 0.71 (0.82) | 1.77 (0.76)

4. Other Pre Specified Outcome: Vaginal Dryness Severity Survey (Individual Analysis)
Description: as for outcome 3
Time Frame: 7 Days
Population: Participants who completed their first week of VR101 use
Measure: Count of Participants; unit: Participants
Groups:
- Improved: Participants whose vaginal dryness severity improved (lower score)
- Same: Participants whose vaginal dryness severity did not change
- Worsened: Participants whose vaginal dryness severity worsened (higher score)
Arm/Group | Improved | Same | Worsened
Number analyzed (Participants) | 66 | 66 | 66
Participants | 48 | 15 | 3

5. Other Pre Specified Outcome: VR101 Ease of Use Survey
Description: Claim 2: VR101 is easy to use by following the provided instructions.
  To assess the ability to use VR101 by following the instructions for use and without professional medical assistance, participants were asked to rate their level of agreement with the following statement, the ring was easy to use by following the provided instructions, when removing their first VR101. The following scale was used to rate the level of agreement:
  * "Disagree completely" (assigned a score of -4)
  * "Disagree a lot" (assigned a score of -3)
  * "Disagree somewhat" (assigned a score of -2)
  * "Disagree a little" (assigned a score of -1)
  * "Neither agree nor disagree" (assigned a score of 0)
  * "Agree a little" (assigned a score of 1)
  * "Agree somewhat" (assigned a score of 2)
  * "Agree a lot" (assigned a score of 3)
  * "Agree completely" (assigned a score of 4)
  The scores of the 67 participants are summarized below. "Favorable" scores were defined as those of 1 or higher.
Time Frame: First Ring Insertion
Measure: Count of Participants; unit: Participants
Groups:
- Favorable: Participants who reported a score of 1 (agree a little) or higher upon inserting their first VR101 device.
- Unfavorable: Participants who reported a score of 0 (neither agree nor disagree) or lower upon inserting their first VR101 device
Arm/Group | Favorable | Unfavorable
Number analyzed (Participants) | 67 | 67
Participants | 62 | 5

6. Other Pre Specified Outcome: Number of VR101 Devices Considered as Comfortable / Uncomfortable
Description: Claim 3: VR101 is comfortable during use
  In each daily diary, the participant was asked to rate her level of agreement with the statement "the ring was comfortable to me today." The following scale was used to rate the level of agreement:
  * "Disagree completely" (assigned a score of -4)
  * "Disagree a lot" (assigned a score of -3)
  * "Disagree somewhat" (assigned a score of -2)
  * "Disagree a little" (assigned a score of -1)
  * "Neither agree nor disagree" (assigned a score of 0)
  * "Agree a little" (assigned a score of 1)
  * "Agree somewhat" (assigned a score of 2)
  * "Agree a lot" (assigned a score of 3)
  * "Agree completely" (assigned a score of 4)
Time Frame: Up to 4 weeks total
Measure: Number; unit: Daily Diary Entries
Groups:
- Favorable: Daily diaries during VR101 use with a comfort score of 1 (agree a little) or higher.
- Unfavorable: Daily diaries during VR101 use with a comfort score of 0 (neither agree nor disagree) or lower.
Arm/Group | Favorable | Unfavorable
Number analyzed (Participants) | 72 | 72
Daily Diary Entries | 1629 | 215

7. Post Hoc Outcome: Efficacy of VR101 Treatments at 28 Days Assessed by Change in VHI (Vaginal Health Index) Scores Assigned by Clinicians - Post-Hoc Analysis 1
Description: The Vaginal Health Index (VHI) ranges from 5 to 20 and is calculated via addition of clinician-determined ratings for Vaginal Elasticity, Fluid Volume, Epithelial Integrity, Moisture and pH (each ranges from 1 to 5, with 5 being the best).
  The SAS Proc Mixed model was employed with Kenward-Roger degrees of freedom. The treatment effect was defined as the change in VHI between baseline and day 28. The subject, sequence, period and treatment were all included as effects. Furthermore, last observation carried forward (LOCF) for the raw score was used for cases where the Day 28 observation was missing within a treatment period if the subject had at least one measurement, including baseline, within the treatment period.
Time Frame: Baseline, 28 Days
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | VR101 | Sham Control
Number analyzed (Participants) | 72 | 72
Score on a Scale
  Baseline Included as Covariate | 1.59 (0.33) | 0.44 (0.34)
  Baseline not included as Covariate | 1.68 (0.41) | 0.35 (0.41)

8. Post Hoc Outcome: Efficacy of VR101 Treatments at 28 Days Assessed by Change in VHI (Vaginal Health Index) Scores Assigned by Clinicians - Post-Hoc Analysis 2
Description: The Vaginal Health Index (VHI) ranges from 5 to 20 and is calculated via addition of clinician-determined ratings for Vaginal Elasticity, Fluid Volume, Epithelial Integrity, Moisture and pH (each ranges from 1 to 5, with 5 being the best).
  The "missingness" of VHI scores was evaluated in detail, with the eventual conclusion that a missing at random (MAR) assumption was plausible for the missing VHI scores (at either day 0 or day 28). This conclusion was supported by the observation that no participants reported withdrawing due to a lack of perceived VR101 efficacy. The analysis also modeled raw VHI values rather than the treatment effect (change in VHI from day 0 to day 28), but reported summary statistics in terms of net treatment effect. No LOCF imputations were performed.
Time Frame: Baseline, 28 Days
Measure: Mean (Standard Error); unit: Score on a Scale
Groups:
- VR101 Net Effect on 28 Day Composite VHI Scores (Adjusted for Sham Control Effect): VR101 Net Effect on 28 day Composite VHI Scores (adjusted for sham control effect)
Arm/Group | VR101 Net Effect on 28 Day Composite VHI Scores (Adjusted for Sham Control Effect)
Number analyzed (Participants) | 72
Score on a Scale
  Classical Mixed Model | 0.48 (0.21)
  Unequal Variance Model | 0.49 (0.20)

ADVERSE EVENTS:
Time Frame: Up to 24 weeks total, including up to 17 weeks total VR101 use and up to 4 weeks total sham use.
Groups:
- VR101: Participants for whom adverse events were reported during VR101 use.
- Sham Control: Participants for whom adverse events were reported during Sham Control use.
Arm/Group | VR101 | Sham Control
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/67
Other Adverse Events (participants affected / at risk) | 46/69 | 31/67
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VR101 (N=69) | Sham Control (N=67)
Inability to remove ring (Product Issues) | 6 | 4
Vaginal Discharge - Mild (Reproductive system and breast disorders) | 2 | 2
Vaginal Discomfort - Mild to Moderate (Reproductive system and breast disorders) | 7 | 3
Increased Urge / Urinary Incontinence - Mild to Moderate (Renal and urinary disorders) | 5 | 2
Vaginal / Labial Bleeding / Spotting [Non-Menstrual] - Mild (Reproductive system and breast disorders) | 4 | 2
Urinary Tract Infection - Mild to Moderate (Renal and urinary disorders) | 3 | 1
Vaginal Itching - Mild (Reproductive system and breast disorders) | 2 | 1
Yeast Infection - Moderate (Reproductive system and breast disorders) | 2 | 0
Abdominal Cramps / Discomfort - Moderate (General disorders) | 1 | 2
Vaginal Burning Sensation - Moderate (Reproductive system and breast disorders) | 1 | 1
Vaginal Bacterial Infection - Moderate (Reproductive system and breast disorders) | 1 | 0
Urethritis - Mild (Renal and urinary disorders) | 1 | 0
Malodor - Mild (Reproductive system and breast disorders) | 1 | 0
Intermittent Nausea - Moderate (General disorders) | 1 | 0
Intermittent Headache - Mild (General disorders) | 1 | 0
Pelvic Pain - Mild (General disorders) | 0 | 1
Vaginal Irritation - Moderate (Reproductive system and breast disorders) | 0 | 1
Excessive Secretions - Mild to Moderate (Reproductive system and breast disorders) | 3 | 0
Other AEs - Not Related to Ring (General disorders) | 35 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT03150407/Prot_SAP_001.pdf